CLINICAL TRIAL: NCT00476268
Title: A 24-week Phase III Study to Evaluate the Efficacy and Tolerability of Beclometasone/Formoterol Single Inhaler HFA 134a-pMDI in Adult Patients With Moderate to Severe Persistent Asthma
Brief Title: Efficacy and Tolerability of Beclometasone/Formoterol Single Inhaler in Patients With Moderate to Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM/PR/033011/003/03
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- beclometasone /formoterol (Experimental): beclomethasone dipropionate 100 µg plus formoterol 6 µg pMDI
  Interventions: Drug: beclomethasone/formoterol (100/6µg) pMDI
- Beclomethasone (Active Comparator): Beclomethasone dipropionate (BecotideTM) 250 µg/unit dose pMDI aerosol via CFC propellant.
  Interventions: Drug: Beclometasone dipropionate 250 µg/unit dose pMDI
- Formoterol powder 12 µg/unit dose (Active Comparator): Formoterol powder 12 µg/unit dose (Foradil™)
  Interventions: Drug: Formoterol powder 12 µg/unit dose

INTERVENTIONS:
Drug: beclomethasone/formoterol (100/6µg) pMDI — Two puffs b.i.d
  Arms: beclometasone /formoterol
Drug: Beclometasone dipropionate 250 µg/unit dose pMDI — 2 inhalations bid
  Other Names: BecotideTM
  Arms: Beclomethasone
Drug: Formoterol powder 12 µg/unit dose — 2 inhalations bid
  Other Names: Foradil™
  Arms: Formoterol powder 12 µg/unit dose

SUMMARY:
Efficacy and tolerability of the fixed combination beclometasone/formoterol in patients with moderate to severe persistent asthma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and tolerability of beclometasone/formoterol single inhaler in a twice daily regimen in patients with moderate to severe persistent asthma. Patients are randomised to receive either beclometasone/formoterol single inhaler (total daily dose: BDP/FF 400/24 mcg) or beclometasone CFC + formoterol DPI (total daily dose: BDP 1000 mcg + FF 24 mcg) or beclometasone CFC (total daily dose: BDP 1000 mcg) during 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe persistent asthma (according to GINA 2002 guidelines)
* FEV1 > 40% and < 80% of predicted normal post-bronchodilator (and at least 0.7 L absolute value)
* Patients already treated for at least 2 months with an association of inhaled corticosteroids plus LABA at doses of:

  750 - 1000 µg beclomethasone dipropionate or equivalent (ICSs) 24 µg formoterol or 100 µg salmeterol (LABAs)
* Or patients naïve of LABA already treated for at least 2 months with inhaled corticosteroids (doses as above) associated with a daily use of SABA and/or with clinical symptoms > 3 times in the week prior to inclusion
* A documented positive response to the reversibility test.

Exclusion Criteria:

* Pregnant or lactating females or women of childbearing potential without any efficient contraception.
* Heavy smokers defined as smoking for > 10 pack years.
* Evidence of asthma exacerbation causing an hospitalisation or requiring treatment with oral/parenteral corticosteroids or evidence of symptomatic airways infection in the 4 weeks prior to inclusion (3 months for slow-release corticosteroids).
* Seasonal asthma or asthma occurring only during episodic exposure to an allergen or occupational chemical sensitizer.
* Clinically significant or unstable concomitant diseases, including clinically significant laboratory abnormalities.
* Patients with an abnormal QTc interval value in the ECG test, defined as > 450 msec in males or > 470 msec in females.
* Evidence of asthma worsening during the week preceding randomisation (e.g. PEF variability > 30% during 2 consecutive days, SABA use > 8 puffs/day during 2 consecutive days, nocturnal awakenings due to asthma symptoms during 3 consecutive days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Actual)
Dates: Start 2004-02; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Pre-dose morning PEF | End of treatment

SECONDARY OUTCOMES:
Pre-dose FEV1 | At clinic visits
Other spirometric parameters | At clinic visits
Morning and evening asthma clinical symptom scores | End of treatment
Percentage of night and/or days free of clinical symptoms | End of treatment
Use of rescue short-acting b2-agonists | End of treatment
Asthma exacerbations | end of treatment
safety and tolerability | end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Bonnet-Gonod, Study Director — Chiesi Farmaceutici

REFERENCES:
- [Result] Huchon G, Magnussen H, Chuchalin A, Dymek L, Gonod FB, Bousquet J. Lung function and asthma control with beclomethasone and formoterol in a single inhaler. Respir Med. 2009 Jan;103(1):41-9. doi: 10.1016/j.rmed.2008.09.002. Epub 2008 Nov 1. PMID 18977646